CLINICAL TRIAL: NCT00226603
Title: Prevention of Groin Injuries in Football Players
Brief Title: Lyske Trial (Danish) Groin Trial
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hölmich, Per, M.D. (Individual)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KF 01-171/97
Record Dates: First submitted 2005-09-23; First posted 2005-09-27 (Estimated); Last update posted 2005-09-27 (Estimated); Status verified 1998-06

CONDITIONS: Groin Injuries in Football Players
Keywords: groin injury; football; prevention; traing programme; cluster randomized study

INTERVENTIONS:
Behavioral: Specific training programme (behavior)

SUMMARY:
To examine the effect of a specific training programme towards groin injuries in male footbal players. To evaluate the effect on other football related injuries as well. To examine any possible relations between various possible predictors such as experience, age, hypermobility and others, and the risk of sustaining inujries during football.

ELIGIBILITY:
Inclusion Criteria:

male adult football players playing in the participating clubs in the study period

-

Exclusion Criteria:

* under 18 years groin injury at the start of the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1600
Dates: Start 1997-09; Study Completion 1998-06

CONTACTS AND LOCATIONS:
Overall Officials: Christian Gluud, PHD, Study Chair — H:S Copenhagen Trial Unit
Locations (1):
- Per Holmich, Copenhagen, Værløse, Denmark